CLINICAL TRIAL: NCT06427603
Title: Sit Less and Move More: A Feasibility Study on Physical Active Break Intervention and Improving Cardiometabolic Health
Brief Title: Sit Less and Move More: Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Bonny WONG Yee Man, Assistant Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD/2022/2.12
Record Dates: First submitted 2024-05-08; First posted 2024-05-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- activity group (Experimental)
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — workshops and mobile apps: break sedentary behavior by activity breaks

SUMMARY:
Intervention aiming to improve cardiometabolic health and physical function by reducing prolonged sitting

ELIGIBILITY:
Inclusion Criteria:

1. are community-dwelling older adults aged 65 years or above,
2. are smartphone users,
3. sit for >= 6 hours per day
4. are overweight

Exclusion Criteria:

1. are unable to walk independently with/without walking aids due to a physical disability;
2. have health conditions that hinder the adherence to intervention

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | T2: post-intervention (week 12)
  will be assessed using a scale "Feasibility, appropriateness, and acceptability of the intervention"

SECONDARY OUTCOMES:
Sedentary behavior | T1: baseline (before the study begins)
  will be assessed using an accelerometer
Sedentary behavior | T2: post-intervention (week 12)
  will be assessed using an accelerometer
Sarcopenia score ranged from 0 to 20 | T1: baseline (before the study begins)
  will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls (SARC-Calf)
Sarcopenia score ranged from 0 to 20 | T2: post-intervention (week 12)
  will be assessed using the Strength, Assistance with walking, Rise from a chair, Climb stairs and (Calf) Falls (SARC-Calf)
Blood glucose | T1: baseline (before the study begins)
  will be assessed using a portable blood monitoring device
Blood glucose | T2: post-intervention (week 12)
  will be assessed using a portable blood monitoring device
Blood pressure | T1: baseline (before the study begins)
  will be assessed using a portable blood monitoring device
Blood pressure | T2: post-intervention (week 12)
  will be assessed using a portable blood monitoring device
Muscle strength (handgrip strength) | T1: baseline (before the study begins)
  will be assessed using a hand-held dynamometer
Muscle strength (handgrip strength) | T2: post-intervention (week 12)
  will be assessed using a hand-held dynamometer
Physical performance | T1: baseline (before the study begins)
  will be assessed using Time-Up-to-Go (TUG)
Physical performance | T2: post-intervention (week 12)
  will be assessed using Time-Up-to-Go (TUG)
physical function | T1: baseline (before the study begins)
  will be assessed using Short physical performance battery (SPPB) ranging 0 to 12
physical function | T2: post-intervention (week 12)
  will be assessed using Short physical performance battery (SPPB) ranging 0 to 12
Physical activity | T1: baseline (before the study begins)
  will be assessed using an accelerometer
Physical activity | T2: post-intervention (week 12)
  will be assessed using an accelerometer
Standing | T1: baseline (before the study begins)
  will be assessed using an accelerometer
Standing | T2: post-intervention (week 12)
  will be assessed using an accelerometer

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing and Health Studies, Hong Kong Metropolitan University, Ho Man Tin, Hong Kong

IPD SHARING:
Plan to Share IPD: No